CLINICAL TRIAL: NCT03836989
Title: Pilot Clinical Trial to Study Facial Electrical Stimulation to Promote Recovery in Patients With Bell's Palsy and Poor Prognostic Factors
Brief Title: Electrical Stimulation to Promote Recovery in Bells Palsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Myriam Loyo, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16901
Record Dates: First submitted 2018-11-19; First posted 2019-02-11 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Bell Palsy
Keywords: Facial Paralysis; Bell Palsy; Electrical Stimulation
MeSH Terms: conditions — Bell Palsy; Facial Paralysis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessors are blinded to the intervention. The physical therapist that teaches the research subjects how to perform the interventions are not blinded and patients are told they are assigned to either sensory or subsensory protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High-volt electrical stimulation (Experimental): Plan to use a monophasic waveform having 100µmsec pulse duration, at 35 Hz using tolerated voltage to generate a contraction a total of 20 minutes.
  The stimulation will have 10 seconds on time, 30 seconds off time and 2 second ramp up and down. Electrical stimulation will be produced with the Orthostim 3 device (VQ Ortho Care). The cathode will be placed on the ipsilateral muscle to stimulate and the anode over the ipsilateral mastoid region.
  Four facial muscles will be stimulated: 1)frontalis, 2) orbicularis oculi, 3) zygomaticus major, and 4) orbicularis oris.
  The voltage is turned up by the participant until he or she can see twitches or as high as tolerated. Ten contractions in each muscle group will be performed or 5 minutes per muscle if no contraction is achieved.
  Interventions: Device: Electrical stimulation device (tens unit)
- Subsensory electrical stimulation (Placebo Comparator): Plan to use the same device and settings to provide placebo treatment by delivering minimal electricity. The settings will be the same as the intervention except the voltage will be subsensory. ie. below the minimum at which patients feels any effect of the current.
  The voltage is turned down two clicks from the voltage at which the participant can first notice any electricity or at the minimal setting.
  Interventions: Device: Electrical stimulation device (tens unit)

INTERVENTIONS:
Device: Electrical stimulation device (tens unit) — An electrical stimulation device with adjustable voltage. Useful for both Sensory and Subsensory

SUMMARY:
A feasibility pilot study to exam the necessary methodology for conducting a larger clinical trial for Bell's Palsy patients with a poor prognosis and the use of electrical stimulation.

DETAILED DESCRIPTION:
Here we describe a protocol for a prospective, randomized, double-blinded study to evaluate the effects of monophasic pulsed current ES on patients with Bell's palsy and factors predicting poor recovery, with a 6 month follow up. Motor level stimulation with a pulse duration of 100 μsec and a frequency of 35 pulses per second were chosen from focus group with physical therapist to treat facial paralysis and are consistent with clinical trials showing motor benefit after capel tunnel surgery.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of bell's palsy (diagnosed in the last 30 days)
* IF younger than 60 years of age must have complete paralysis on one side of face or both
* IF older than 60 years of age paralysis must be present but CAN be incomplete.

Exclusion Criteria:

* Paralysis associated with any of the fallowing: cancer, tumor, surgery, stroke, or trauma.
* Younger than 60 years old with INCOMPLETE paralysis.
* Non English speakers
* Pacemaker or deep brain stimulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myriam D Loyo, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Blocks were designed to account for predictors of recovery. There were four allocation blocks: 1) >60 age with complete paralysis, 2) > 60 age with incomplete paralysis, 3) <60 age with complete paralysis and < 15 days duration, or 4) <60 age with complete paralysis and >15 days duration.
  The block size was 2 and the allocation was 1:1. All patients were randomly allocated to high-volt arm
Period: Overall Study
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Started | 4 | 0
Subjects > 60 Years Old With Complete Paralysis | 1 | 0
Subjects > 60 Years Old With Incomplete Paralysis | 1 | 0
Subject < 60 Years Old + Complete Paralysis < 15 Days Duration | 1 | 0
Subjects < 60 Years Old + Complete Paralysis > 15 Days | 1 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomization led to no participants in the Subsensory arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 1 |  | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Recovery at 3 Months as Measured From Facial Photos With Different Facial Expressions
Description: To evaluate for complete recovery, standardized photos of patients at rest, and during movement, will be evaluated by three treatment-blinded otolaryngologists. Total number of patients fully recovered over number of participants will be reported.
Time Frame: 3 months
Population: Randomization led to no Subsensory participants.
Measure: Count of Participants; unit: Participants
Groups:
- High-volt Electrical Stimulation: Plan to use a monophasic waveform having 100µmsec pulse duration, 35 Hz and using tolerated voltage for a total of 20 minutes. Electrical stimulation will be produced with the Orthostim 3 device. The cathode will be placed on the ipsilateral muscle to stimulate and the anode over the ipsilateral arm.
  The voltage is turned up by the participant until he or she can see twitches or as high as tolerated.
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
Participants | 3 |

2. Secondary Outcome: House Brackmann Scale
Description: Determined by three blinded otolaryngologist reviewing facial photos of patients with smile and eye closure. Reported as an average of the three scores. The scales ranges from 1 (normal) to 6 (most severe dysfunction)
Time Frame: Baseline, and 3 months
Population: No subjects underwent subsensory electrical stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High-volt Electrical Stimulation: Plan to use a monophasic waveform having 100µmsec pulse duration, at 35 Hz using tolerated voltage to generate a contraction a total of 20 minutes.
  The stimulation will have 10 seconds on time, 30 seconds off time and 2 second ramp up and down. Electrical stimulation will be produced with the Orthostim 3 device (VQ Ortho Care). The cathode will be placed on the ipsilateral muscle to stimulate and the anode over the ipsilateral mastoid region.
  Four facial muscles will be stimulated: 1)frontalis, 2) orbicularis oculi, 3) zygomaticus major, and 4) orbicularis oris.
  The voltage is turned up by the participant until he or she can see twitches or as high as tolerated. Ten contractions in each muscle group will be performed or 5 minutes per muscle if no contraction is achieved.
  Electrical stimulation device (tens unit): An electrical stimulation device with adjustable voltage. Useful for both Sensory and Subsensory
- Subsensory Electrical Stimulation: Plan to use the same device and settings to provide placebo treatment by delivering minimal electricity. The settings will be the same as the intervention except the voltage will be subsensory. ie. below the minimum at which patients feels any effect of the current.
  The voltage is turned down two clicks from the voltage at which the participant can first notice any electricity or at the minimal setting.
  Electrical stimulation device (tens unit): An electrical stimulation device with adjustable voltage. Useful for both Sensory and Subsensory
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
score on a scale
  3 months | 2 (1.15) |
  Baseline | 5.5 (1) |

3. Secondary Outcome: Patient Reported Quality of Life in Relation to Facial Synkinesis Measured by the Synkinesis Assessment Questionnaire (SAQ)
Description: Quality of life is in part measured in this study using the patient reported Synkinesis Assessment Questionnaire (SAQ). The instrument consisting of 10 items asks participants how difficult certain facial activities are. Based on the average score for each domain the test gives a score between 20 (no synkinesis) to 100 (severe synkinesis, all the time).
Time Frame: Baseline, 3 months and 6 months
Population: No research subjects participated in the subsensory electrical stimulation arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
score on a scale
  3 month outcome | 27.5 (5.25) |
  6 month outcome | 38.7 (23.5) |
  Baseline | 31 (7.7) |

4. Secondary Outcome: Patient Reported Global Quality of Life Specific to Facial Paralysis
Description: Measured by the validated quality of life patient reported questionnaire Facial Clinimetric Evaluation (FaCE) Scale with a scale from 0 (normal) to 100 (severe dysfunction). The scale encompasses facial movement, facial comfort, oral function, eye comfort, lacrimal control, and social function.
Time Frame: Baseline, 3 months and 6 months
Population: No subjects were recruited for the subsensory arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
score on a scale
  Baseline | 37.5 (3.4) |
  3 months | 51.25 (12.03) |
  6 months | 51 (15) |

5. Secondary Outcome: Objective Measurements of Brow Elevation
Description: Measuring brow elevation using the MEEI FACE-gram program reported as the millimeters in decreased elevation in comparison to the unaffected side
Time Frame: Baseline and in 3 months
Population: No subjects were allocated to the subsensory arm
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
millimeters
  Baseline | 7.75 (2.2) |
  3 months | 4.5 (5.2) |

6. Secondary Outcome: Eye Closure
Description: Measuring in millimeters of the eyelids remaining open during maximal eye closure using the MEEI FACE-gram program
Time Frame: Baseline and 3 months
Population: No subjects were allocated to the subsensory arm
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
millimeters
  Baseline | 2.5 (3.1) |
  3 months | 0.5 (0.6) |

7. Secondary Outcome: Smile Excursion
Description: Measuring oral commissure exclusion using the MEEI FACE-gram program reported as the change in millimeters in the distance between the midline of the lower lip and the oral commissure in comparison between rest and smile
Time Frame: Baseline and 3 months
Population: No subjects were allocated to the subsensory arm
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
millimeters
  Baseline | -1 (1.15) |
  3 months | 4.5 (3.5) |

8. Secondary Outcome: Facial Symmetry at Rest
Description: Measured by facial asymmetry index (FAI) at rest in photos which is calculated as the difference in the distance from the lateral canthus to the oral commissure between the affected and unaffected side. In the scale 0 equals no difference between sides and perfect symmetry. The closer a number is to 0, the higher the symmetry is. Ranges have not been published for this scale. FAI does not have a maximum score.
Time Frame: Baseline and 3 months
Population: No subjects were allocated to the subsensory arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
score on a scale
  Baseline | 0.25 (0.2) |
  3 months | 0.02 (0) |

9. Secondary Outcome: Facial Symmetry During Smile
Description: Measured by facial asymmetry index (FAI) during smile in photos which is calculated as the difference in the distance from the lateral canthus to the oral commissure between the affected and unaffected side. In the scale 0 equals perfect symmetry and no difference in sides. The closer a number is to 0, the greater the symmetry. Ranges have not been published for this scale. FAI does not have a maximum score.
Time Frame: Baseline and 3 months
Population: no subjects were allocated to the subsensory arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
score on a scale
  Baseline | 0.4 (0.6) |
  3 months | 0.2 (0.19) |

10. Secondary Outcome: Patient Tolerability
Description: Measured by a visual analog scale (VAS) which ranged from 0 to 10 where 0 stands for completely comfortable and 10 to very uncomfortable. A questionnaire designed by research team using a Likert's scale was created to measure patient tolerability.
Time Frame: 3 months
Population: No subjected were recruited for the subsensory arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
score on a scale | 2.7 (2.3) |

11. Secondary Outcome: Self Reported Subject Adherence
Description: Percentage of subjected who reported full adherence, partial adherence and non-adherence confirmed by comparing to the daily diary of use.
Time Frame: 3 months
Population: no subjects were recruited to the subsensory electrical stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | High-volt Electrical Stimulation | Subsensory Electrical Stimulation
Number analyzed (Participants) | 4 | 0
Participants
  Full adherence | 4 |
  Partial adherence | 0 |
  Non adherence | 0 |

ADVERSE EVENTS:
Time Frame: Adverse event data will be collected throughout the participants therapy. Therapy is to start during the first week of onset of facial paralysis and be used daily for three months or sooner until complete recovery is achieved. Adverse event data was collected for up to 3 months
Description: No participants were enrolled in the subsensory stimulation.
Groups:
- High-volt Electric Stimulation: Plan to use a monophasic waveform having 100µmsec pulse duration, at 35 Hz using tolerated voltage to generate a contraction a total of 20 minutes.
  The stimulation will have 10 seconds on time, 30 seconds off time and 2 second ramp up and down. Electrical stimulation will be produced with the Orthostim 3 device (VQ Ortho Care). The cathode will be placed on the ipsilateral muscle to stimulate and the anode over the ipsilateral mastoid region.
  Four facial muscles will be stimulated: 1)frontalis, 2) orbicularis oculi, 3) zygomaticus major, and 4) orbicularis oris.
  The voltage is turned up by the participant until he or she can see twitches or as high as tolerated. Ten contractions in each muscle group will be performed or 5 minutes per muscle if no contraction is achieved
- Subsensory Electric Stimulation: Plan to use the same device and settings to provide placebo treatment by delivering minimal electricity. The settings will be the same as the intervention except the voltage will be subsensory. ie. below the minimum at which patients feels any effect of the current.
  The voltage is turned down two clicks from the voltage at which the participant can first notice any electricity or at the minimal setting.
Arm/Group | High-volt Electric Stimulation | Subsensory Electric Stimulation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 3/4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-volt Electric Stimulation (N=4) | Subsensory Electric Stimulation (N=0)
Pain (Nervous system disorders) | 1 (1) | 0
Headache (Nervous system disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT03836989/Prot_SAP_000.pdf